CLINICAL TRIAL: NCT05447611
Title: Role of Empathy in the Outcome of Curative Treatment of Non-metastatic Colorectal Cancer. Prospective Multicenter Longitudinal Study in Two Departments Covered by the Calvados Cancer Registry.
Brief Title: Role of Empathy in Curative Treatment Outcomes of Non-metastatic Colorectal Cancer.
Acronym: EMPACOL
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Other Study IDs: 22-0065
Record Dates: First submitted 2022-06-21; First posted 2022-07-07 (Actual); Last update posted 2022-07-07 (Actual); Status verified 2022-06

CONDITIONS: Non-metastatic Colorectal Cancer; Empathy; Morbidity; Morality; Quality of Life
Keywords: colorectal cancer; empathy; outcomes
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- high score CARE group: Patient-perceived empathy was assessed using the Consultation and Relational Empathy (CARE) questionnaire that has been validated in cancer care. This is a self-reported ten-point questionnaire with a five-point Likert-type scale ranging from "poor" to "excellent" Likert-type scale. It has excellent psychometric properties with α = 0.92. High scores indicate a higher perception of the health care personnel empathy.
  The three distinct empathic processes were also assessed with the CARE measure. 'Relationship' was assessed with items 1-3, 'emotional process' with items 4-6, and 'cognitive process' with items 7-10.
- lower score CARE group: In line with the recent literature, we considered differentiating the study population into two groups: those with a high perceived empathy (maximum CARE score) and those without.

SUMMARY:
The aim of project EMPACOL will be to investigate, while taking into consideration the clinical factors known and well described in the literature, among the non-clinical factors, in particular, patient-healthcare personnel (HCP) relationship, a link between HCP's empathy perceived by the patient, and the results of the curative treatment of non-metastatic colorectal cancer, throughout the patient's care.

DETAILED DESCRIPTION:
EMPACOL will be a multicenter prospective longitudinal study. Over a 2-year period, in two French areas covered by a cancer register, 8 centers will include patients with non-metastatic CRC, uncomplicated at diagnosis Based on the curative treatment strategy, patients will be divided into three groups: group 1 (surgery alone), group 2 (surgery and adjuvant chemotherapy), group 3 (neo-adjuvant therapy, surgery and adjuvant chemotherapy).

The relationship between HCP's empathy, perceived by the patient, after 2 years of inclusion, and the quality of life (QoL) at one year after the end of treatment will be investigated. QoL will be investigated using the QLQ C-30 questionnaire. Finally, a link between PHC perception and oncological outcomes will be sought.

ELIGIBILITY:
Inclusion Criteria:

Patients aged 18 to 75 years, French-speaking, affiliated to a social security system, having received informed information and not having expressed an unfavorable opinion to participate; carriers of non-metastatic and uncomplicated CRC (without occlusion/ perforation/bleeding), requiring elective therapeutic management. The included patients have a cognitive state capable of understanding and completing the questionnaires (autonomous completion).

Exclusion Criteria:

Patients who were minors or older than 80 years, residing in a department outside Calvados or Manche, presenting a CRC other than adenocarcinoma and all metastatic forms or requiring emergency surgery (perforation, hemorrhage, occlusion), exclusive endoscopic treatment, or a missed-CRC discovered after surgery for non-oncological indications.

Patients with another neoplastic disease under treatment and/or evolving, patients with a history of inflammatory bowel disease (Crohn's disease, ulcerative colitis) and/or hereditary disease predisposing to CRC (Lynch syndrome, familial polyposis) or with severe cognitive impairment preventing proper comprehension of the questionnaires. Pregnant women will be excluded.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Medical information included gender, age, obesity, active smoking and alcohol use alcohol , the ASA physical status classification system (I-II versus III-IV), anxious and depressive states (HADS score) of patient and presentation at multidisciplinary consultation, histology and tumor differentiation, surgical approach, as well as neoadjuvant or adjuvant treatments (type and number of sessions), site of the primary tumor (colon vs rectum). The forms located at the rectosigmoid junction were included in the colonic localizations.
  All patients diagnosed with CRC during the inclusion period were included in two specialized digestive cancer registries of North-West France, members of the French network of cancer registries (FRANCIM), department of Calvados and Manche.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2022-09 (Estimated); Primary Completion 2024-09 (Estimated); Study Completion 2029-09 (Estimated)

PRIMARY OUTCOMES:
The main objective of the EMPACOL project is to investigate, in non-metastatic CRC patients, a possible correlation, between perceived HCP's empathy and survival (OS and DFS). | 5 years of follow up
  Based on the curative treatment strategy, patients with non-metastatic CRC will be divided into three groups: group 1 (surgery alone), group 2 (surgery and adjuvant chemotherapy), group 3 (neo-adjuvant therapy, surgery and adjuvant chemotherapy).
  The relationship between patient-perceived HCP empathy after 2 years of inclusion and 5-year survival will be studied.

SECONDARY OUTCOMES:
The relationship between caregiver empathy, as perceived by the patient, and quality of life (QoL) will be studied. | One year after the end of treatment
  Quality of life will be studied using the QLQ C-30 questionnaire.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mulliri A, Lelorain S, Bouvier V, Bara S, Gardy J, Grynberg D, Morello R, Alves A, Dejardin O. Role of empathy in the outcomes of colorectal cancer: protocol for a population-based study in two areas in France (EMPACOL Project). BMJ Open. 2022 Nov 29;12(11):e066559. doi: 10.1136/bmjopen-2022-066559. PMID 36446452